CLINICAL TRIAL: NCT00522080
Title: Screening for Hip and Knee Osteoarthritis in the General Population: Predictive Value of a Questionnaire and Prevalence Estimates
Status: Terminated | Type: Observational
Why Stopped: terminated study
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Other Study IDs: 04-CIR-07
Record Dates: First submitted 2007-08-27; First posted 2007-08-29 (Estimated); Last update posted 2007-08-29 (Estimated); Status verified 2007-08

CONDITIONS: Hip and Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Time Perspective: Other
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Objective: To study the feasibility and validity of a two-step telephone screening procedure for symptomatic knee and hip osteoarthritis (OA) in the general population.

Method: The screening questionnaire was based on signs and symptoms, previous diagnosis of OA, and validated OA criteria. A random sample of telephone numbers was obtained and, at each number, one individual aged 40 to 75 years was included. A physical examination and knee or hip radiographs were offered when the screen was positive. A sample of individuals with negative screens was also examined. The diagnosis of hip/knee OA was based on either American College of Rheumatology criteria for signs and symptoms and Kellgren-Lawrence radiographic stage 2 or greater. Prevalence rates were estimated with correction for the performance of the screening procedure.

ELIGIBILITY:
Inclusion Criteria:

* Individual aged 40 to 75 years

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Dates: Start 2005-03; Study Completion 2005-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: christian h roux, Dr, Principal Investigator — CHU NICE
Locations (1):
- Rheumatology department, Nice University hospital, Nice, France